CLINICAL TRIAL: NCT00952237
Title: Immune Mobilization of Autologous Peripheral Blood Stem Cells Using Interleukin-2 and GM-CSF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Meehan, Director, Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0227
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2016-05

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma; Other Plasma Cell Dyscrasia (Waldenstrom, Amyloidosis); Leukemia
Keywords: Autologous Peripheral Blood Stem Cell Transplant; IL-2; GM-CSF
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Amyloidosis; Leukemia | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IL-2 and GM-CSF for Mobilization (Experimental): Immune Mobilization of Autologous Peripheral Blood Stem Cells Using Interleukin-2 and GM-CSF
  Interventions: Drug: GM-CSF; Drug: IL-2

INTERVENTIONS:
Drug: GM-CSF — GM-CSF (Recombinant Human Granulocyte-Macrophage Colony Stimulating Factor) The dose and duration of GM-CSF (7.5 mcg/kg/day) was selected. If used alone, this dose and duration would result in effective mobilization. GM-CSF will be started on Day #7 and will continue until completion of leukapheresis.
  G-CSF will be started (5mcg/kg/d) on Day #7 and will be given each morning. G-CSF will continue until completion of leukapheresis.
Drug: IL-2 — IL-2 dose escalation: IL-2 will be administered as a single daily subcutaneous injection each evening until completion of leukapheresis.
  Escalation of the dose of IL-2 will be performed using the below schema with the following levels. Patients will be started on Level 1. (Level 0 is included since, if toxicity is meet in Level 1, the dose will be decreased to Level 0).
  Level 0 - 3 x 105 i.u./m2/day for 11 days Level 1 - 6 x 105 i.u./m2/day for 11 days Level 2 - 1 x 106 i.u. /m2/day for 11 days as above Level 3 - 1.5 x 106 i.u. /m2/day for 11 days as above Level 4 - 2 x 106 i.u. /m2/day for 11 days as above

SUMMARY:
We postulate that the combination of IL-2 and GM-CSF immunotherapy will efficiently mobilize autologous peripheral blood stem cells and activated immune effector cells in patients with a hematologic malignancy. These activated effector cells will improve the immune function of the graft. These hypotheses will be tested using this proposed clinical trial to mobilize autologous peripheral blood stem cells pre-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have pathologic diagnosis of one of the following malignancies: Non-Hodgkin's Lymphoma, Hodgkin's Disease, Multiple Myeloma or other plasma cell dyscrasia (Waldenstrom, Amyloidosis), Leukemia (AML, ALL, CLL)
* Prior Treatment: > 2 weeks prior to initiation of therapy.
* Performance Status: Karnofsky > 70%
* Age >18
* Life Expectancy > 4 months
* Bone Marrow: bone marrow biopsy and aspirate
* Blood counts: The patient must have adequate bone marrow function, i.e. a total WBC of > 2,000/ul, a Hgb of > 7 mg/dl, and a platelet count of > 50,000/ul, unless this abnormality is believed to be due to the underlying disease.
* Pulmonary function tests: DLCO > 55% predicted.
* Cardiac: Left ventricular ejection fraction of > 40% by radionuclide scan or echocardiography.
* Liver function tests (bilirubin, alkaline phosphatase, and SGOT/SGPT) < 3 x normal (unless believed to be elevated due to disease).
* No significant co-morbid medical or psychiatric illness that would significantly compromise the patient's clinical care and chances of survival.
* Informed Consent: Informed consent must be signed prior to the treatment. Patients must be aware of the neoplastic nature of their disease and willingly consent after being informed of the procedure to be followed, the nature of the therapy, alternatives, potential benefits, side effects, risks and discomforts. The patient is not deemed eligible if there is any other serious medical or psychiatric illness that would prevent informed consent. (Human protection committee approval of this protocol and a consent form is required.)

Exclusion Criteria:

* Medical, social, or psychological factors which would prevent the patient from receiving or cooperating with the full course of therapy.
* Evidence on physical exam, LP, CT, or MRI scans of CNS involvement with malignancy.
* Uncontrolled or severe cardiovascular disease, including recent (< 6 months) myocardial infarction, congestive heart failure, angina (symptomatic despite optimal medical management), life-threatening arrhythmia, or hypertension or clinically significant obstructive/restrictive pulmonary disease.
* Serology positive for HIV
* History of seizures.
* Concurrent or expected need for therapy with systemic corticosteroids (since systemic steroids may suppress the effects of IL-2).
* Current and clinically significant pleural effusion, pericardial effusion, or ascites.
* Positive pregnancy test or presence of lactation.
* Uncontrolled active infection.
* Documented hypersensitivity to any of the drugs used in the protocol.
* No concomitant, ongoing malignancy that is life-threatening, based on PI's evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Can IL-2 be administered with GM-CSF to efficiently mobilize autologous peripheral blood stem cells. This study will determine the maximum tolerated dose of IL-2 and the optimal biological dose with GM-CSF for stem cell mobilization. | 5 Years

SECONDARY OUTCOMES:
Will immune-mobilized stem cell products be well tolerated once infused into patients and will engraft normally following high-dose chemotherapy and APBSCT. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Meehan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States